CLINICAL TRIAL: NCT02957032
Title: A Dose-finding Phase I Study of the Tumor-targeting Human F16IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Very Low-dose Cytarabine in Patients With AML Relapse After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: A Study of the Tumor-targeting Human F16IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Very Low-dose Cytarabine in Patients With AML Relapse After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New agents for the same indication impacted on patients' recruitment
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-F16IL2CYT-03/14
Record Dates: First submitted 2016-10-17; First posted 2016-11-07 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acute Myeloid Leukemia, Relapsed, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Cytarabine

ARMS (1):
- F16IL2 + cytarabine (Experimental): Patients will be enrolled sequentially in cohorts and treated at different dose levels of F16IL2 and a fixed dose of cytarabine.
  Interventions: Drug: F16IL2; Drug: cytarabine

INTERVENTIONS:
Drug: F16IL2 — All patients first receive an initial run-in dose of 30 Mio IU of F16IL2 on day 1 and escalating doses of F16IL2 on day 1, 8, 15 and 22.
  Treatment will be repeated every 28 days for up to three cycles.
Drug: cytarabine — Patients will be treated with cytarabine (5 mg twice daily s.c. for 10 days). Treatment will be repeated every 28 days for up to three cycles.

SUMMARY:
Phase I, open label, non-randomized, multicenter, prospective dose escalation study of F16IL2 in combination with very low-dose cytarabine in subjects with acute myeloid leukemia relapse after allogeneic hematopoietic stem cell transplantation (alloHSCT).

DETAILED DESCRIPTION:
Phase I, open label, non-randomized, multicenter, prospective dose escalation study of F16IL2 in combination with very low-dose cytarabine in subjects with acute myeloid leukemia relapse after allogeneic hematopoietic stem cell transplantation (alloHSCT).

The aim of the study is to determine a recommended dose for F16IL2 in AML relapse after alloHSCT and investigating the toxicity of the combination regimen.

Patients will be enrolled sequentially in cohorts and treated at different dose levels of F16IL2 and a fixed dose of cytarabine. All patients first receive an initial run-in dose of 30 Mio IU of F16IL2 on day 1 and escalating doses of F16IL2 on day 1, 8, 15 and 22. Patients will be treated with cytarabine (5 mg twice daily s.c. for 10 days). The following F16IL2 administration will be at the dose of the respective cohort (days 8, 15 and 22).

The RD will be defined following a traditional 3+3 design. The dose escalation will continue until the MTD is found, that is until at least two patients among a cohort of three to six patients experience a dose limiting toxicity (DLT) (i.e., >33 % of patients with a DLT). The RD is defined as the dose level just below the MTD level. If the MTD is not found at cohort 5 the RD for this study will be considered equal to the cohort 5 dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML (except APL) relapse after alloHSCT meeting the following criteria (at least one feature must be present):

   * bone marrow blasts ≥ 5% of all nucleated cells
   * appearance of blasts in the peripheral blood
   * extramedullary AML relapse.
2. Age ≥18 years.
3. ECOG ≤ 2.
4. Documented negative test HIV-HBV-HCV. For HBV serology: the determination of HBsAg, anti-HBsAg-Ab and anti-HBCAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required.
5. Negative serum pregnancy test for females of childbearing potential* within 14 days of starting treatment.
6. Informed consent, personally signed and dated to participate in the study.
7. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

   * Women of childbearing potential (WOCBP) must be using, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesteron-only or combined (estrogen- and progesteron-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomised partner or sexual abstinence. Pregnancy test will be repeated at the end of treatment visit.

Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilised (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

Exclusion Criteria:

1. Known central nervous system manifestation of AML.
2. Previous therapy (chemotherapy, radiotherapy, investigational drugs) for this current AML relapse after alloHSCT, unless this previous treatment yielded in a documented progression of the disease and except hydroxyurea to control peripheral cell counts up to 24h before study medication.
3. Active GvHD requiring systemic immunosuppression, unless controlled with low dose steroids equivalent to a maximum of 10 mg methylprednisolone per day.
4. All acute toxic effects of any prior therapy returned to G≤1 according to CTCAE v4.03 (excluding alopecia)
5. Chronically impaired renal function (creatinine clearance < 30 ml/min).
6. Inadequate liver function (ALT, AST, AP or total bilirubin ≥ 3.0 x ULN), if not caused by leukemic infiltration.
7. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
8. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
9. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
10. Irreversible cardiac arrhythmias requiring permanent medication.
11. LVEF < 50%
12. Uncontrolled hypertension.
13. Ischemic peripheral vascular disease (Grade IIb-IV). Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
14. Major trauma including surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
15. Pregnancy or breast feeding.
16. Requirement of chronic administration of corticosteroids. However, low dose corticosteroids (maximum 10 mg methylprednisolone (or equivalent) per day when administered for GVHD or cancer symptoms (e.g., pain, dyspnoea, lack of appetite).
17. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
18. Known active or latent tuberculosis (TB).
19. Concurrent malignancies other than AML (except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the patient has been disease-free for at least 2 years.
20. Concomitant treatment with angiogenesis inhibitors or other drugs with proven anti-leukemic activity.
21. Serious, non-healing wound, ulcer or bone fracture.
22. Allergy to study medication or excipients in study medication (not including drug fever or rash to cytarabine).
23. Concurrent use of other anti-cancer treatments or agents with the exception of palliative radiation, e.g. to myelosarcoma lesions not blinding the efficacy judgement of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04-13 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Safety assessment will be performed from Day 1 up to Day 28 of the Cycle 1 (each cycle is 28 days)
  To assess the safety, including maximum tolerated dose (MTD), recommended dose (RD) and dose limiting toxicity (DLT) of F16IL2 combined with very low dose cytarabine, Adverse Events (AEs) assessment based on CTCAE v.4.03 will be considered.

SECONDARY OUTCOMES:
The overall response rate (ORR, consisting of CR and CRi as defined by the International Working Group (IWG) criteria). | Up to 13 months
The relapse-free survival (RFS) of responding (CR and CRi) patients. | Up to 12 months
The time to response (CR or CRi) of responding patients. | Up to 13 months
Median progression free survival (PFS) | Up to 13 months
Median overall survival (OS) | Up to 13 months
The time to complete donor chimerism. | Up to 13 months
The rate to complete donor chimerism. | Up to 13 months
The rate of acute GvHD. | Up to 13 months
The rate of chronic GvHD. | Up to 13 months
  The rate of patients with chronic GvHD will be summarized according to the following Chronic GVHD Staging:
  * mild: involvement of 1 to 2 organs/sites (except for lung) with a maximum score of 1;
  * moderate: involvement of at least 1 organ/site with a score of 2 or ≥ 3 organs/sites with a score of 1 or lung involvement with a score of 1;
  * severe: any organ/site with a score of 3 or lung involvement with a score of 2.
Human anti-fusion protein antibodies (HAFA) levels before and following treatment. | at Day 1 (cycle 1), at Day 29 (cycle 2), Day 57 (cycle 3), from Day 25 to Day 85 (EoT visit), from Day 53 to Day 113 (first follow-up visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Münster University Hospital, Münster, Germany